CLINICAL TRIAL: NCT06742957
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multiple-Site, Clinical Study to Evaluate the Therapeutic Equivalence of Tapinarof Cream 1% (Teva Pharmaceuticals, Inc.) With VTAMA® Tapinarof (Tapinarof) Cream 1% (Dermavant Sciences, Inc.) in Adult Patients With Plaque Psoriasis
Brief Title: Study Comparing Tapinarof Cream 1% To VTAMA ® (Tapinarof Cream 1%) In the Treatment of Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Collaborators: Teva Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 72336004
Record Dates: First submitted 2024-12-16; First posted 2024-12-19 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Plaque Type Psorisis
Keywords: Dermatologic Agents; Skin Diseases; Plaque Psoriasis; Tapinarof; Adult; Phase 3; Topical; Double-Blind; Safety; Efficacy; Skin Diseases, Papulosquamous
MeSH Terms: conditions — Skin Diseases; Skin Diseases, Papulosquamous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Test: Tapinarof Cream 1% (Experimental): Tapinarof Cream 1%, Apply a thin layer once daily to psoriatic affected areas for 84 days.
  Interventions: Drug: Tapinarof Cream 1%
- VTAMA® (Active Comparator): (Tapinarof) Cream 1%, Apply a thin layer once daily to psoriatic affected areas for 84 days.
  Interventions: Drug: VTAMA®
- Vehicle Product (Placebo Comparator): Vehicle of the Test Product, Cream, Apply a thin layer once daily to psoriatic affected areas for 84 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tapinarof Cream 1% — Cream
  Arms: Test: Tapinarof Cream 1%
Drug: VTAMA® — Cream
  Arms: VTAMA®
Drug: Placebo — Cream
  Arms: Vehicle Product

SUMMARY:
To compare the safety and efficacy of the test (Tapinarof Cream 1%), placebo (vehicle cream) and reference VTAMA® (Tapinarof Cream 1%) treatments to demonstrate clinical equivalence in patients with plaque psoriasis.

DETAILED DESCRIPTION:
To compare the safety of Test, Reference, and Placebo treatments in patients with Plaque Psoriasis. Patients in this randomized, double-blind, three-arm, placebo controlled, parallel-design, multi-site study will be randomly assigned in a 2:2:1 ratio to treatment with the test product, reference product or placebo control, respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Signed ICF indicating that the patient understands the purpose of, and procedures required for the study and is willing to participate in the study.
2. Males and non-pregnant, non-lactating females aged ≥18 at the time of signing the informed consent.
3. Patients with clinical diagnosis of chronic plaque psoriasis and stable disease for at least 6 months prior to the study.
4. Body surface area (BSA) involvement ≥ 3% and ≤ 20% (the patient's face, scalp, groins, palms and soles should be excluded from the percent of total BSA (%BSA) calculations).
5. A Physician's Global Assessment (PGA) score of 2 (mild), 3 (moderate) or 4 (severe) at screening and baseline.
6. Female patients of childbearing potential (*WOCBP) must not be pregnant or lactating at the time of screening/baseline visit as documented by a negative urine pregnancy test with a sensitivity to at least 25 mIU/ml hCG:

   *Female patients of childbearing potential (WOCBP) are defined as sexually mature women without prior hysterectomy, or who have had any evidence of menses in the past 12 months. However, women who have been amenorrheic for the past 12 or more months are still considered to be of childbearing potential, if the amenorrhea is possibly due to other causes, including prior chemotherapy, anti- estrogens, or ovarian suppression. Postmenopausal women (defined as women who have been amenorrheic for at least 12 consecutive months, in the appropriate age group, without other known or suspected primary cause) or women who have been sterilized surgically or who are otherwise proven sterile (i.e., total hysterectomy, or bilateral oophorectomy with surgery at least 4 weeks prior to randomization) are not considered WOCBP. Patients who have undergone tubal ligation are NOT considered as surgically sterile.
7. Female patients of childbearing potential must be willing to use an acceptable form of birth control during the study from the day of the first dose administration to 30 days after the last administration of study drug.

   1. For the purposes of this study the following are considered acceptable methods of birth control: oral or injectable contraceptives, contraceptive patches, medroxyprogesterone acetate (ex. Depo-Provera®) with stabilized use for at least 3 months, vaginal contraceptive (ex. etonogestrel/ethinyl estradiol vaginal ring (ex. NuvaRing®), contraceptive implant with etonogestrel or equivalent, double barrier methods, (e.g. condom and spermicide), intrauterine device (IUD), true abstinence (if in line with patient's lifestyle).
   2. Patients on hormonal contraception must be stabilized on the same type for at least three months prior to enrollment in the study and must not change the method during the study. A sterile sexual partner is not considered an adequate form of birth control.
   3. If a patient who was abstinent becomes sexually active during the study, a second acceptable method of birth control should be used and documented.
8. Willing and able to adhere to the lifestyle restrictions specified in this protocol.
9. Patients must be in good health and free from any clinically significant disease, which may interfere with the evaluation of plaque psoriasis or the administration of the investigative product.
10. Patients must be willing to refrain from using all other topical plaque psoriasis products during the 12-week treatment period, other than the investigational product.

Exclusion Criteria:

1. Known allergies, hypersensitivity, or intolerance to any of the ingredients of study treatment interventions, or components/ excipients thereof (refer to the prescribing information of VTAMA®), or drug or other allergy that, in the opinion of the investigator, contraindicates participation in the study.
2. Current diagnosis of unstable forms of psoriasis (other than plaque variant) in the treatment area, including guttate, erythrodermic, exfoliative or pustular psoriasis.
3. Patients with other inflammatory skin disease in the treatment area that may confound the evaluation of the plaque psoriasis (e.g., atopic dermatitis, contact dermatitis, tinea corporis, and or any others in the opinion of the Investigator).
4. Presence of pigmentation, extensive scarring, or pigmented lesions in the treatment areas, which could interfere with the rating of efficacy parameters.
5. Patients with current immunosuppression.
6. Ultraviolet (UV) light therapy or prolonged exposure to natural or artificial sources of UV radiation (eg, phototherapy, tanning booths, or therapeutic sunbathing), laser therapy, tattoos removal, skin wraps or exfoliant techniques or Fraxel within 4 weeks prior to the baseline visit and/or plans to have such exposures during the study which could potentially impact the patient's psoriasis (as determined by the Investigator).
7. Use of biological treatments for psoriasis within the last 6 months of the baseline evaluation.
8. Patients that have been treated with systemic steroids, systemic antibiotics, systemic anti-psoriatic treatment (i.e., methotrexate, cyclosporine, hydroxyurea), PUVA therapy, ultraviolet- B Therapy or systemic anti-inflammatory agents within 1 month or within 5 half-lives (whichever is longer) before Baseline.
9. Use of any of the following therapies within two weeks prior to baseline:

   * topical anti-psoriatic drugs (e.g., salicylic acid, anthralin, coal tar, calcipotriene, tazarotene)
   * topical corticosteroids
   * immunosuppressive drugs (e.g., tacrolimus, pimecrolimus)
   * topical retinoids
10. Received an investigational intervention within 30 days or 5 half-lives prior to the first dose of study intervention, whichever is longer.
11. Documented medical history of uncontrolled, clinically significant intercurrent medical condition(s) (i.e., chronic infectious disease, system disorder, organ disorder, cardiovascular, gastrointestinal, hematological, hepatic, neurological, pancreatic, renal disease, severe psychiatric condition, etc.) for which, in the opinion of the investigator, participation would not be in the best interest of the patient (e.g., compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments.
12. Employees of the Investigator or research center or their immediate family members.
13. Females who are pregnant, breast feeding, or who wish to become pregnant during the study period.
14. Patients who have received chemotherapy or radiation therapy and/or anti-neoplastic agents within 3 months prior to screening/baseline.
15. Patients who are unable or unwilling to give informed consent.
16. Patients, who in the opinion of the Investigator, would be non-compliant with the requirements of the study protocol.
17. Patients who consume excessive amounts of alcohol (greater than two drinks per day) or use drugs of abuse (including, but not limited to, cannabinoids, cocaine and barbiturates) within one year prior to screening.
18. Patients who have been previously enrolled in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 560 (Actual)
Dates: Start 2024-12-17 (Actual); Primary Completion 2025-10-07 (Actual); Study Completion 2025-11-12 (Actual)

PRIMARY OUTCOMES:
Primary change in the Physician Global Assessment (PGA) | 12 Weeks
  Proportion of patients with treatment success (defined as a Physician Global Assessment (PGA) score of clear (0) or almost clear (1) with a minimum 2-grade improvement from baseline at the end of treatment (Week 12; Study Day 84):
  Score of (0) Clear: No signs of psoriasis; post-inflammatory hyperpigmentation may be present
  Score of (1) Almost Clear: No thickening; normal to pink coloration; no to minimal focal scaling
  Score of (2) Mild: Just detectable to mild thickening; pink to light red coloration; predominantly fine scaling
  Score of (3) Moderate: Clearly distinguishable to moderate thickening; dull to bright red, clearly distinguishable erythema; moderate scaling
  Score of (4) Severe: Severe thickening with hard edges; bright to deep dark red coloration; severe/coarse scaling covering almost all or all lesions

CONTACTS AND LOCATIONS:
Locations (26):
- United States (26):
  - Site 12107, Scottsdale, Arizona
  - Site 12101, Bryant, Arkansas
  - Site 12110, Dublin, California
  - Site 12112, Dublin, California
  - Site 12102, Fremont, California
  - Site 12119, Huntington Beach, California
  - Site 12120, Northridge, California
  - Site 12111, Pomona, California
  - Site 12122, Greenwich, Connecticut
  - Site 12115, Fort Lauderdale, Florida
  - Site 12104, Miami, Florida
  - Site 12116, Miami, Florida
  - Site 12113, Miami, Florida
  - Site 12114, Miramar, Florida
  - Site 12108, Chicago, Illinois
  - Site 12121, Rolling Meadows, Illinois
  - Site 12106, Clarksville, Indiana
  - Site 12123, Merrillville, Indiana
  - Site 12105, Louisville, Kentucky
  - Site 12109, Las Vegas, Nevada
  - 12127, Woodbury, New York
  - Site 12126, Portland, Oregon
  - Site 12125, Upper Saint Clair, Pennsylvania
  - Site 12103, College Station, Texas
  - Site 12118, El Paso, Texas
  - Site 12117, Houston, Texas

REFERENCES:
- See also: FDA Drug and Device Resources — https://clinicaltrials.gov/fda-links
- See also: Office of Generic Drugs, Center for Drug Evaluation and Research. Draft Guidance on Tapinarof (PSG_215272) [Internet]. Silver Spring, MD: U.S. Food and Drug Administration; 2023 [cited 2024 May 10]. — https://www.accessdata.fda.gov/drugsatfda_docs/psg/PSG_215272.pdf
- See also: VTAMA (Tapinarof) cream, 1%, for topical use [US Prescribing Information] [Internet]. Long Beach, CA: Dermavant Sciences Inc.; 2023 [cited 2024 May 16]. — https://dailymed.nlm.nih.gov/dailymed/drugInfo.cfm?setid=9309d20f-8cd4-4c96-93fa-7f730e83c7ab